CLINICAL TRIAL: NCT05914376
Title: A Phase I Dose Escalation Study to Evaluate the Safety, Tolerance, Pharmacokinetics, and Biological Properties of Recombinant Human IL-21-expressing Oncolytic Vaccinia Virus Injection (hV01) in Patients With Advanced Malignant Solid Tumors
Brief Title: Safety of Recombinant Human IL-21-expressing Oncolytic Vaccinia Virus Injection (hV01) in Advanced Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Converd Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: hV01-ITu-101
Record Dates: First submitted 2023-05-31; First posted 2023-06-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hV01 intratumoral injection (Experimental): Single-dose phase (3+3 design):
  Participants will receive an intratumoral injection of hV01 at one of the dose levels from 1.0×10^7 PFU to 8.0×10^8 PFU on Day 1 of each treatment cycle. The MTD or MAD will be determined based on the safety and tolerability outcomes of this phase.
  Multiple-dose phase (3+3 design):
  1. Two doses per cycle: Participants will receive two intratumoral injections of hV01 at the dose level of sub-MTD or sub-MAD on Day 1 and Day 8 of each treatment cycle.
  2. Three doses per cycle: Participants will receive three intratumoral injections of hV01 at the dose level of sub-MTD or sub-MAD on Day 1, Day 8 and Day 15 of each treatment cycle.
  Interventions: Biological: Recombinant human IL-21-expressing oncolytic vaccinia virus injection

INTERVENTIONS:
Biological: Recombinant human IL-21-expressing oncolytic vaccinia virus injection — hV01 is a recombinant vaccinia virus with deletions of the viral thymidine kinase (TK) and viral growth factor (VGF) genes and insertion of the human IL-21 gene.
  Other Names: hV01

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerance, pharmacokinetics, and biological properties of recombinant human IL-21-expressing oncolytic vaccinia virus injection (hV01) in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multi-site, single-arm, open-label, dose-escalation study. It consists of two phases: Part A involves a single-dose escalation, and Part B evaluates the safety and tolerability of multiple doses of hV01.

Part A: Dose escalation with four dose levels from 1.0×10^7 PFU to 8.0×10^8 PFU. The standard 3+3 dose escalation design will be used to determine the maximum tolerated dose (MTD) or maximum administered dose (MAD). The participants will be observed for dose-limiting toxicities (DLTs) for 28 days after the single dose of the first cycle.

Part B: After completion of Part A, the sub-MTD/MAD will be chosen for Part B, which will evaluate the safety and tolerability of hV01 administration at two different frequencies: twice per cycle (on days 1 and 8) and three times per cycle (on days 1, 8, and 15). The standard 3+3 design will also be used for this phase. The first cohort, receiving two doses per cycle, will be observed for DLTs for 35 days after the first dose, while the second cohort, receiving three doses per cycle, will be observed for DLTs for 42 days after the first dose.

ELIGIBILITY:
Inclusion Criteria:

* Signing an informed consent form.
* Men or women aged 18 to 75 years.
* Histologically and/or cytologically confirmed advanced malignant solid tumors refractory or failed to respond to standard therapy (including disease progression and/or intolerable toxicities).
* At least one measurable lesion according to RECIST v1.1 criteria, which can be injected intratumorally either directly or with the assistance of medical imaging equipment such as B-ultrasound or CT. The baseline longest diameter (shortest diameter for lymph node lesions) of the lesion targeted for injection should be more than 1.5 cm, and the lesion also meets the requirements of the relevant dosing volume.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Life expectancy of at least 3 months.
* Required baseline laboratory data include:

  1. Hematology: absolute neutrophil count (ANC) ≥ 1.5×10^9/L, platelet (PLT) count ≥ 75×10^9/L, hemoglobin (Hb) ≥90 g/L (without supportive therapy within 14 days prior to laboratory test);
  2. Liver function: serum total bilirubin (TBIL) ≤1.5×ULN (or ≤3×ULN for patients with Gilbert's syndrome or liver metastasis); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3×ULN (or<5×ULN for patients with primary liver cancer or liver metastasis);
  3. Renal function: serum creatinine (Cr) ≤1.5×ULN, and creatinine clearance (Cockcroft-Gault method) ≥45 mL/min. For men: creatinine clearance = [[140-age(yr)]×weight (kg)]/[0.818×creatinine (μmol/L)]; For women: creatinine clearance = [[140-age(yr)]×weight (kg)×0.85]/[0.818×creatinine (μmol/L)];
  4. Coagulation test: activated partial thromboplastin time (APTT) ≤1.5×ULN; international normalized ratio (INR) ≤1.5×ULN.
* Female patients of childbearing age must have a negative serum pregnancy test. Female patients of childbearing age and male patients whose partners are of childbearing age must agree to use medically approved contraceptive measures (hormonal or barrier methods or abstinence) throughout the treatment period and also within 3 months after the last dose of the investigational drug. Male patients must also avoid sperm donation.

Exclusion Criteria:

* Receiving any of the following anti-tumor treatments within a specified time period:

  1. Systemic anti-tumor treatment, including chemotherapy, large-molecule targeted therapy, immunotherapy, and endocrine therapy within 4 weeks before first dose (within 6 weeks of dosing for nitrosourea or mitomycin C);
  2. Small-molecule targeted therapy within 2 weeks before first dose or within 5 half-lives of the small-molecule targeted drug (whichever is longer);
  3. Traditional Chinese medicine or Chinese herbal medicine used as anti-tumor agent within 2 weeks before first dose;
  4. Radiotherapy (excluding palliative radiotherapy) within 2 weeks before first dose;
  5. Prior oncolytic virus treatment.
* Acute toxic effects from prior treatments not resolved to Common Terminology Criteria for Adverse Events (CTCAE, v5.0) grade 1 or below, except for toxicities deemed safe by the investigator, such as alopecia.
* Patients with clinical symptoms of central nervous system (CNS) metastasis or meningeal metastasis, or other evidence indicating that CNS or meningeal metastases are not controlled.
* Known or suspected active autoimmune diseases (including but not limited to systemic lupus erythematosus, Sjogren's syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, and Hashimoto's thyroiditis).
* Previous allogeneic stem cell or organ transplantation.
* History of severe cardiovascular and cerebrovascular diseases, including:

  1. Acute coronary syndrome (including myocardial infarction, severe or unstable angina), myocarditis, congestive heart failure, cerebrovascular accidents, or other cardiovascular events of CTCAE (v5.0) grade 3 or higher within 12 months of dosing;
  2. Severe arrhythmia requiring clinical intervention (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes), corrected QT interval (QTc) >450 ms for males or >470 ms for females, or a family history of long QT syndrome;
  3. New York Heart Association (NYHA) classification of class II or above, or left ventricular ejection fraction (LVEF) <50%;
  4. Uncontrolled hypertension (as judged by the investigator) or hypotension despite standard treatment.
* Any uncontrolled active infection requiring systemic anti-infective therapy (graded 2 or higher according to CTCAE v5.0), including but not limited to active tuberculosis, sepsis, bacteremia, fungemia, and viremia.
* Any of the following infections: human immunodeficiency virus (HIV), syphilis spirochete(TP), active hepatitis C (positive HCV RNA test) or active hepatitis B (positive HBsAg and HBV DNA ≥ 2000 IU/mL or ≥10^4 copies/mL).
* Use of immunomodulatory drugs within 2 weeks of dosing, including but not limited to thymosin, interleukin, interferon.
* Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2025-10-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
To assess the Dose-limiting toxicities (DLTs) of hV01. | From first dose till 28 days after last dose.
  To identify dose-limiting toxicities (DLTs) of hV01 administered by single or multiple intratumoral injections.
To assess the adverse events (AEs) and tolerability of hV01. | From informed consent to approximately 3 months after End of Trial (EOT)
  To assess the frequency, severity, and nature of adverse events (AEs) of hV01 administered by single or multiple intratumoral injections at different dose levels. This will be determined by abnormalities or changes in vital signs, Eastern Cooperative Oncology Group (ECOG) performance status, physical examination, 12-lead electrocardiogram, and laboratory test results.

SECONDARY OUTCOMES:
Pharmacokinetics of hV01. | From baseline to 28 days after last dose.
  To evaluate the hV01 DNA concentrations in peripheral blood at different time points.
Expression of IL-21. | From baseline to 28 days after last dose.
  To evaluate IL-21 levels in peripheral blood at different time points.
Viral shedding of hV01. | From baseline to 28 days after last dose.
  To evaluate hV01 DNA levels in urine and feces, and also quantities of hV01 DNA recovered from throat swab and injection site swab.
Anti-tumor activity of hV01: overall response rate (ORR). | From baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years after the end of treatment.
  To evaluate the overall response rate (ORR) as a measurement of tumor response and disease progression.
Anti-tumor activity of hV01: disease control rate (DCR). | From baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years after the end of treatment.
  To evaluate the disease control rate (DCR) as a measurement of tumor response and disease progression.
Anti-tumor activity of hV01: duration of response (DOR). | From baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years after the end of treatment.
  To evaluate the duration of response (DOR) as a measurement of tumor response and disease progression.
Anti-tumor activity of hV01: progression-free survival (PFS). | From baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years after the end of treatment.
  To evaluate the progression-free survival (PFS) as a measurement of tumor response and disease progression.
Preliminary efficacy of hV01: overall survival (OS). | From signing informed consent form until the date of death from any cause, assessed up to 2 years after the end of treatment.
  To evaluate the overall survival (OS) as a measurement of preliminary efficacy.

OTHER OUTCOMES:
To evaluate the immunogenicity of hV01. | From baseline to 4 weeks after the End of Treatment.
  To assess the levels of anti-drug antibody (ADA) and neutralizing antibody (Nab) in the peripheral blood.
To assess immune cells in the peripheral blood | From baseline to 4 weeks after the End of Treatment.
  To assess the levels of lymphocytes (CD3+ cells, CD3+CD4+ cells, CD3+CD8+ cells, CD3+CD4+/CD3+CD8+, CD3-CD16+CD56+ cells, CD3-CD19+ cells) in the peripheral blood.
To assess cytokine levels in the peripheral blood. | From baseline to 4 weeks after the End of Treatment.
  To assess the levels of cytokines including IFN-γ, TNF-α, and IL-6 in the peripheral blood.
To assess the correlation between anti-tumor responses and expressions of tumor biomarkers | From baseline until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years after the end of treatment.
  To assess the impact of baseline Epidermal Growth Factor Receptor (EGFR) or Vascular Endothelial Growth Factor Receptor (VEGFR) mutation on tumor response after hV01 treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Zhejiang People's Hospital, Hangzhou, Zhejiang
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No